CLINICAL TRIAL: NCT06849544
Title: Phase II Trial to Investigate the Safety and Efficacy of Four Dosing Regimens of OTL78 Injection (Zopocianine), a Prostate-Specific Membrane Antigen (PSMA)-Targeted Fluorescent Agent, for the Intraoperative Imaging of Prostate Cancer
Brief Title: Phase II Trial to Investigate the Safety and Efficacy of Four Dosing Regimens of OTL78 Injection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinton Bahler (Other)
Collaborators: Indiana University Melvin and Bren Simon Cancer Center (Other); On Target Laboratories, LLC (Industry)
Responsible Party: Sponsor-Investigator, Clinton Bahler, Associate Professor, Indiana University
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UROL-CC-IUSCCC-0902
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer Surgery; Prostate Cancer Metastatic Disease
Keywords: Prostate Specific Membrane Antigen; Fluorescent Imaging; Near infrared imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 0.03mg/kg ZOPOCIANINE given day of surgery (Experimental): A single dose of 0.03mg/kg ZOPOCIANINE (given 1 - 12 hours prior to surgery) used with NIR fluorescent imaging during prostatectomy and lymph node dissection for biopsy confirmed prostate cancer.
  Interventions: Drug: 0.03mg/kg ZOPOCIANINE given day of surgery
- 0.06mg/kg ZOPOCIANINE given day prior to surgery (Experimental): A single dose of 0.06mg/kg ZOPOCIANINE (given 12 - 30 hours prior to surgery) used with NIR fluorescent imaging during prostatectomy and lymph node dissection for biopsy confirmed prostate cancer.
  Interventions: Drug: 0.06mg/kg ZOPOCIANINE given day of surgery
- 0.03mg/kg ZOPOCIANINE given day prior to surgery (Experimental): A single dose of 0.03mg/kg ZOPOCIANINE (given 12 - 30 hours prior to surgery) used with NIR fluorescent imaging during prostatectomy and lymph node dissection for biopsy confirmed prostate cancer.
  Interventions: Drug: 0.03mg/kg ZOPOCIANINE given day prior to surgery
- 0.06mg/kg ZOPOCIANINE given 2-7 days prior to surgery (Experimental): A single dose of 0.06mg/kg ZOPOCIANINE (given 2-7 days prior to surgery) used with NIR fluorescent imaging during prostatectomy and lymph node dissection for biopsy confirmed prostate cancer.
  Interventions: Drug: 0.06mg/kg ZOPOCIANINE given days prior to surgery

INTERVENTIONS:
Drug: 0.03mg/kg ZOPOCIANINE given day of surgery — A single dose of 0.03mg/kg ZOPOCIANINE used with NIR fluorescent imaging during prostatectomy and lymph node dissection
  Arms: 0.03mg/kg ZOPOCIANINE given day of surgery
Drug: 0.06mg/kg ZOPOCIANINE given day of surgery — A single dose of 0.06mg/kg ZOPOCIANINE used with NIR fluorescent imaging during prostatectomy and lymph node dissection
  Arms: 0.06mg/kg ZOPOCIANINE given day prior to surgery
Drug: 0.03mg/kg ZOPOCIANINE given day prior to surgery — A single dose of 0.03mg/kg ZOPOCIANINE used with NIR fluorescent imaging during prostatectomy and lymph node dissection
  Arms: 0.03mg/kg ZOPOCIANINE given day prior to surgery
Drug: 0.06mg/kg ZOPOCIANINE given days prior to surgery — A single dose of 0.06mg/kg ZOPOCIANINE used with NIR fluorescent imaging during prostatectomy and lymph node dissection
  Arms: 0.06mg/kg ZOPOCIANINE given 2-7 days prior to surgery

SUMMARY:
This study is being done to compare how well Zopocianine (OTL78) in combination with Near InfraRed (NIR) fluorescent imaging may improve the detection of malignant (growing in an uncontrolled way) tissue in adult subjects undergoing prostatectomy and lymph node dissection for biopsy confirmed prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the second leading cause of cancer-related death behind lung cancer. Prostate cells express Prostate Specific Membrane Antigen (PSMA), which is overexpressed in PCa cells in over 90% of patients. On Target has developed a PSMA-targeted agent, the drug product OTL78, that fluoresces under NIR illumination to help with the identification of prostate cancer tissue during resection surgery that has extended beyond the capsule of the prostate into adjacent tissue and lymph nodes. Intra-operative identification of cancer tissue using real-time imaging modalities that could improve tumor identification, demarcation and lymph node involvement may provide a very useful tool to reduce the frequency of residual cancer and increase complete removal of locally involved lymph nodes. This study is an open label trial of an imaging agent, PSMA targeted fluorescent dye (zopocianine, OTL78), in up to 20 subjects with biopsy confirmed PCa who have been scheduled to undergo a laparoscopic radical prostatectomy with pelvic lymph node dissection in order to explore the relationship between the amount of drug given, the timing of administration relative to surgery, and the utility of the drug in visualizing cancerous tissue during a standard of care radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent and HIPAA form
2. Male subjects 18 years of age and older
3. Known primary prostate cancer and Grade Group 3 to 5 (≥ cT3) or one or more of the following:

   1. Suspected extraprostatic disease (EPD) (extracapsular extension (ECE) and/or seminal vesicle infiltration (SVI)),
   2. 3 or more biopsy cores of grade group 3-5;
   3. Suspected lymph node metastasis (clinical stage cN1, or by magnetic resonance imaging (mriN+), or by Prostate Specific Membrane Antigen positron emission tomography (PSMA PET+));
4. Planned to undergo a standard of care robotic prostatectomy and lymph node dissection
5. Ability to understand the requirements of the study and agree to abide by the study restrictions and to return for the required assessments
6. Agree to use a medically acceptable method of birth control (e.g., spermicide in conjunction with a barrier such as a condom) or sexual abstinence for the duration of the study, including through final study visit (6 weeks) after the dose of study drug. Sperm donation is prohibited during the study and for 3 months after the dose of study drug. Female partners must use hormonal or barrier contraception unless postmenopausal or abstinent.

Exclusion Criteria:

1. The surgeon plans to perform an extraperitoneal approach
2. History of anaphylactic reactions to products containing indocyanine green
3. History of allergy to any of the components of ZOPOCIANINE:

   1. 2-[3-(1,3-dicarboxypropyl)ureido] pentanedioic acid (DUPA)
   2. Polyethylene glycol-dipeptide linker
   3. Chlorodye
4. Impaired renal or hepatic function:

   1. Renal: creatinine clearance (eGFR) < 50 mL/min
   2. Hepatic: total bilirubin > 2 × upper limit of normal or ALT/AST > 3 × upper limit of normal.
5. Patients with QTc interval ≥ 470 msec per electrocardiogram (ECG) at screening.
6. Significant acute or chronic medical, neurologic, or illness in the subject that, in the judgment of the Principal Investigator, could compromise subject safety, limit the ability to complete the study, and/or compromise the objectives of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 19 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Porportion of subjects who have a Clinically Significant Event | Day of surgery
  1. Histologically confirmed cancer in residual non-nodal soft tissue resected solely because of "NIR only" detection as suspicious following prostatectomy.
  2. One or more resected NIR- positive lymph nodes that contain metastatic disease as confirmed by pathology.

SECONDARY OUTCOMES:
Detection of Primary cancer | Day of surgery
  For primary cancer, the number of lesions that are either: fluorescence positive, and prostate cancer positive (i.e., true positive); fluorescence positive but cancer negative (i.e., false positive); fluorescence negative but cancer positive (i.e., false negative); or, fluorescence negative and cancer negative (i.e., true negative). We will consider disease state at four (4) defined prostate regions - right posterior, left posterior, anterior, and at the bladder neck
Detection of Metastatic Cancer | Day of surgery
  For metastatic cancer spread to lymph nodes, the number of lesions that are either: fluorescence positive, and prostate cancer positive (i.e., true positive); fluorescence positive but cancer negative (i.e., false positive); fluorescence negative but cancer positive (i.e., false negative); or, fluorescence negative and cancer negative (i.e., true negative). We will use six (6) defined lymph node regions (external iliac, internal iliac, common iliac and right and left).
Execution of pre-surgery plan | Day of surgery
  The pre-surgery plan will be documented and compared to the documented surgery performed if surgeon reports of changes in scope from initial plan.
Safety and tolerability of ZOPOCIANINE | Screening to 6 week follow-up
  Incidence rates of all causally related AEs and all SAEs

OTHER OUTCOMES:
Cancer detected by NIR only | Day of Surgery
  Number of tissues that are fluorescence positive and histologically confirmed cancer which were not detected by pre-operative PSMA-PET scanning.

CONTACTS AND LOCATIONS:
Overall Officials: Clint Bahler, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Indiana University Health North Hospital, Carmel, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes